CLINICAL TRIAL: NCT06241053
Title: Effects of Multimodal Physical Therapy With and Without McConnell Taping in Patients With Anterior Knee Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0148
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Anterior Knee Pain; McConnell taping; Patellofemoral Pain Syndrome.
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Combined Modality Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants of both groups will be informed about the possible risks and potential.
  benefits but they won't know which group they are placed in. The participants must sign consent forms agreeing to the experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal therapy with McConnell taping (Experimental): Multimodal therapy includes core exercises, hip exercises and vastus medialis training.
  MacConnell taping will be applied during exercise and then nearly for 18 hours according to patient's comfort.
  Interventions: Other: Multimodal therapy with McConnell taping
- Multimodal therapy without McConnell taping (Experimental): Multimodal therapy includes core exercises, hip exercises and vastus medialis training.
  Interventions: Other: Multimodal therapy without McConnell taping

INTERVENTIONS:
Other: Multimodal therapy with McConnell taping — Multimodal therapy includes core exercises, hip exercises and vastus medialis training.
  Core exercises include curls ups, toa taps, side planks, supine straight leg raising, side lying straight leg raising, prone knee flexion, draw foot circles in supine and side lying, prone cobra, hip and knee extension, weight bearing, hip flexion sitting on ball, wight bearing forward and backward on the ball, stairs up on Swiss ball. Hip training includes Hip abduction, Hip external rotation in standing and sitting. VMO muscle strengthening will includes squats with a ball.
  Arms: Multimodal therapy with McConnell taping
Other: Multimodal therapy without McConnell taping — Multimodal therapy without McConnell taping
  Arms: Multimodal therapy without McConnell taping

SUMMARY:
This study aims to determine the effect Multimodal physical therapy with and without McConnell taping on pain, functional limitation and severity of symptoms in patients with anterior knee pain.

DETAILED DESCRIPTION:
The term "Anterior Knee Pain" is often used interchangeably with "Patellelofemoral Pain Syndrome" (PFPS or " runner's knee" which involves stiffness and pain when patellofemoral joint is loaded with different activities that require prolonged knee flexion, stairs climbing or descending , running, kneeling and squatting. Multimodal therapy and tapping techniques are useful for reducing pain and improving functional activities of patient daily living.

In this randomized clinical trial, Thirty participants with anterior knee pain will be randomly assigned to one of the two intervention groups: Group A: Group A will be treated with multimodal physical therapy program with McConnell taping. Group B: Group B will be treated with multimodal physical therapy program without McConnell taping. Randomization will be performed using a convenient random sampling method via lottery method. Each participant will receive a total of 12 treatment sessions.

over a four-week period. The effects of the interventions will be assessed at the beginning (first session), conclusion (eight session). Participants will be followed up after 4 weeks again. Outcome measures, including pain intensity, functional limitation and severity of symptoms will be evaluating using the Visual Analog Scale (VAS), Lower Extremity Functional Scale (LEFS) and Anterior Knee Pain Scale (AKPS) respectively. Data will be analyzed using SPSS software version 25. Normality of data will be assessed using the Shapiro-wilk test. For within-group comparisons, paired t- test will be used. To compare changes between the groups, the independent t-test will be applied, depending on the data distribution. The analysis of these outcome measures will provide. valuable insights into the impact of the interventions on participants' pain, functional limitation and severity of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 17-35 years, both male and female.
* Unilateral or bilateral pain lasting for more than 2-3 months.
* Diagnosed with patellofemoral pain by orthopedic surgeon through clinical and radiological findings.
* Positive patellofemoral grinding test, negative McCurry test and full knee range of motion.
* Pain grade 3-6 by Visual Analogue Scale (VAS).
* Pain at least in two of these positions: sitting for long time with knee bends, going up and down the stairs, squatting and running, kneeling.

Exclusion Criteria:

* History of ligament sprain, meniscal injury, knee fracture, patellar dislocation and knee osteoarthritis.
* True knee joint locking or giving away and tibial or iliotibial track tendinopathy.

Pregnancy.

* Developmental dysplasia of hip and undergoing any medical treatment.
* Spinal surgery and neurological disorders.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-02-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 4rth week
  Visual analog scale is a self-assessing questionnaire comprising 10cm line with 0 representing no pain and 10 is worst pain. Reliability of VAS in patients with anterior knee pain is .60 to .79 for usual pain and .88 for worst pain.
Lower Extremity Functional Scale | 4rth week
  The Lower Extremity Functional Scale is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The score for each task is separated in 5 categories "0" (extreme difficulty or unable to perform activity), "1" (quite a bit of difficulty), "2" (moderate difficulty), "3" (a little bit of difficulty) and "4" (no difficulty). The maximal function is 80 points.
Anterior Knee Pain Scale | 4rth week
  The Anterior Knee pain Scale questionnaire consist of 13 items assessing subjective symptoms and functional limitation of the patients with anterior knee pain. The score ranges from 0 (worst condition) to 100 (normal knee condition, no symptoms and no daily functional restrictions).

CONTACTS AND LOCATIONS:
Overall Officials: Ahtsam Liaqat, Principal Investigator — Riphah International University
Locations (1):
- Usman Srawr, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foroughi F, Sobhani S, Yoosefinejad AK, Motealleh A. Added Value of Isolated Core Postural Control Training on Knee Pain and Function in Women With Patellofemoral Pain Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Feb;100(2):220-229. doi: 10.1016/j.apmr.2018.08.180. Epub 2018 Sep 26. PMID 30267667
- [Background] Motealleh A, Kordi Yoosefinejad A, Ghoddosi M, Azhdari N, Pirouzi S. Trunk postural control during unstable sitting differs between patients with patellofemoral pain syndrome and healthy people: A cross-sectional study. Knee. 2019 Jan;26(1):26-32. doi: 10.1016/j.knee.2018.10.002. Epub 2018 Nov 22. PMID 30472048